CLINICAL TRIAL: NCT00841763
Title: A Phase III, Randomized, Controlled, Observer-blind, Multicenter Study to Evaluate the Safety, Tolerability and Immunogenicity of Two Doses of a Monovalent A/H5N1 Influenza Vaccine Adjuvanted With MF59 (Fluad-H5N1) in Adult and Elderly Subjects
Brief Title: Safety, Tolerability and Immunogenicity of Two Doses of Adjuvanted Monovalent Influenza Vaccine Administered to Healthy Adult and Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V87P13; 2008-003871-32 (EudraCT Number)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2019-08

CONDITIONS: Pandemic Influenza Disease
Keywords: virus; pandemic influenza; vaccine
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIV + aH5N1 (Experimental): First dose of the non-adjuvanted trivalent influenza virus vaccine (TIV) followed by two doses of the adjuvanted monovalent influenza virus vaccine (aH5N1).
  Interventions: Biological: Trivalent influenza virus vaccine (TIV); Biological: Adjuvanted monovalent influenza virus vaccine (aH5N1)
- PL + aTIV (Active Comparator): First dose of placebo (PL-saline) followed by two doses of the adjuvanted trivalent influenza virus vaccine (aTIV).
  Interventions: Biological: Placebo (PL); Biological: Adjuvanted trivalent influenza virus vaccine (aTIV)

INTERVENTIONS:
Biological: Placebo (PL) — One dose of 0.5 ml IM injection of isotonic saline solution was administered in the deltoid muscle, preferably of the non-dominant arm.
  Arms: PL + aTIV
Biological: Trivalent influenza virus vaccine (TIV) — A single IM injection of a 0.5 ml dose of non-adjuvanted trivalent influenza virus vaccine administered in the deltoid muscle, preferably of the non-dominant arm.
  Arms: TIV + aH5N1
Biological: Adjuvanted monovalent influenza virus vaccine (aH5N1) — Two intramuscular (IM) injections of a 0.5 ml dose administered three weeks apart in the deltoid muscle.
  Arms: TIV + aH5N1
Biological: Adjuvanted trivalent influenza virus vaccine (aTIV) — Two IM injections of a 0.5 ml dose of adjuvanted trivalent influenza virus vaccine administered three weeks apart, in the deltoid muscle.
  Arms: PL + aTIV

SUMMARY:
The present study, phase III, randomized, controlled, observer-blind, multicenter study, will evaluate safety, tolerability and immunogenicity of two doses of an adjuvanted monovalent influenza vaccine compared with an adjuvanted interpandemic trivalent influenza vaccine in a population of healthy adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age and older who were mentally competent and who had signed an informed consent form after having received a detailed explanation of the study protocol;
* In good health as determined by:

  1. medical history,
  2. physical examination,
  3. clinical judgment of the Investigator;
* Able to understand and comply with all study procedures and to complete study diaries, could be contacted, and were available for study visits;

Exclusion Criteria:

* Receipt of another investigational agent within 4 weeks;
* Laboratory-confirmed influenza disease within 6 months prior to Visit 1;
* Receipt of influenza vaccination for current season 2008/2009;
* Experienced any acute disease or infection requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis was acceptable) within the past 7 days;
* Experienced fever (defined as axillary temperature ≥38.0°C) within 7 days prior to Visit 1;
* Pregnant or breastfeeding;
* Females of childbearing potential who were sexually active and had not used or did not plan or refused to use an acceptable method of birth control during the active phase of the study (at least up to three weeks after last vaccine injection);
* Any serious disease, such as: cancer, autoimmune disease (including rheumatoid arthritis); diabetes mellitus type I and type II; diabetes relating to genetic defects/syndromes, diseases of the exocrine pancreas or infections; advanced arteriosclerotic disease; severe chronic obstructive pulmonary disease (COPD), i.e. GOLD stages 3 and 4; acute or progressive hepatic disease and renal disease; congestive heart failure; Body Mass Index (BMI) ≥35 kg/m2 where BMI reflects obesity and not high muscle mass;
* History of progressive or severe neurologic disorders, of any neurological symptoms or signs, or anaphylactic shock following administration of any study vaccine;
* Bleeding diathesis;
* Surgery planned during the study period;
* Hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the study vaccines;
* Known or suspected impairment/alteration of immune function, for example, resulting from:

  1. receipt of immunosuppressive therapy (any corticosteroid therapy or cancer chemotherapy) or other immunosuppressive agents within the past 60 days and for the full length of the study;
  2. receipt of immunostimulants;
  3. receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study;
  4. suspected or known HIV infection or HIV-related disease;
* Receipt of non study vaccines (with the exception of post-exposure vaccination in a medical emergency, e.g. hepatitis, rabies, tetanus) within 3 weeks prior to Visit 1 or planned vaccination within 3 weeks following the last study vaccination;
* History of (or current) drug or alcohol abuse that in the investigator's opinion would interfere with safety of the subject or the evaluation of study objectives;
* Members of research staff and their relatives;
* Any condition, which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3647 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Director — Novartis Vaccines
Locations (2):
- Tampere Vaccine Research Clinic (15 sites), Tampere, Finland
- 12 Sites, München, Germany

REFERENCES:
- [Result] Vesikari T, Forsten A, Herbinger KH, Cioppa GD, Beygo J, Borkowski A, Groth N, Bennati M, von Sonnenburg F. Safety and immunogenicity of an MF59((R))-adjuvanted A/H5N1 pre-pandemic influenza vaccine in adults and the elderly. Vaccine. 2012 Feb 8;30(7):1388-96. doi: 10.1016/j.vaccine.2011.12.009. Epub 2011 Dec 20. PMID 22192847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 27 centers across Finland and Germany.
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- TIV + aH5N1 (18-60 Yrs): First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
- PL+ aTIV (18-60 Yrs); PL+ aTIV (>60 Yrs): First dose of placebo (PL) followed by two doses of adjuvanted seasonal trivalent influenza vaccine (aTIV).
- TIV + aH5N1 (>60 Yrs): First dose of non adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 influenza vaccine (aH5N1).
Period: Overall Study
Arm/Group | TIV + aH5N1 (18-60 Yrs) | PL+ aTIV (18-60 Yrs) | TIV + aH5N1 (>60 Yrs) | PL+ aTIV (>60 Yrs)
Started | 2691 | 681 | 219 | 56
Completed | 2529 | 624 | 211 | 53
Not Completed | 162 | 57 | 8 | 3
Not completed — Withdrawal by Subject | 60 | 17 | 4 | 1
Not completed — Adverse Event | 9 | 10 | 3 | 2
Not completed — Lost to Follow-up | 63 | 25 | 0 | 0
Not completed — Protocol Violation | 20 | 3 | 1 | 0
Not completed — Administrative Reasons | 3 | 1 | 0 | 0
Not completed — Unable to Classify | 7 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The enrolled set as randomized is reported in the Participant Flow Module but in the Baseline Measure module, the enrolled set as treated is reported (2 randomization errors, 2 subjects were changed from TIV + aH5N1 group to PL+ aTIV group). Moreover, a subset to the enrolled population as treated excluded the one subject who was not vaccinated.
Groups:
- TIV + aH5N1: First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
- PL+ aTIV: First dose of placebo (PL) followed by two doses of adjuvanted seasonal trivalent influenza vaccine (aTIV).
- Total: Total of all reporting groups
Arm/Group | TIV + aH5N1 | PL+ aTIV | Total
Number analyzed (Participants) | 2911 | 735 | 3646
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: Subjects analyzed is not consistent with Participant module due to randomization errors.
  Years
    <= 60 years: number analyzed (Participants) | 2692 | 679 | 3371
    <= 60 years | 40.7 (11.6) | 40.5 (12.0) | 40.7 (11.7)
    >60 years: number analyzed (Participants) | 219 | 56 | 275
    >60 years | 61.9 (1.4) | 62.1 (1.8) | 61.9 (1.5)
Sex/Gender, Customized [Number; unit: participants] — Population: The enrolled set as randomized is reported in the Participant Flow Module but in the Baseline Measure module, the enrolled set as treated is reported (2 randomization errors, 2 subjects were changed from TIV + aH5N1 group to PL+ aTIV group). Moreover, a subset to the enrolled population as treated excluded the one subject who was not vaccinated.
  participants
    Female (<=60 yrs) | 1502 | 388 | 1890
    Male (<=60 yrs) | 1190 | 291 | 1481
    Female (>60 yrs) | 109 | 28 | 137
    Male (>60 yrs) | 110 | 28 | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Reactogenicity Sign After Two Doses of the Adjuvanted Pandemic Influenza Vaccine.
Description: To assess the safety and tolerability profile of two doses of the MF59-adjuvanted A/Vietnam/1194/2004 pandemic influenza vaccine (aH5N1), each containing 7.5 μg of H5N1 antigen in terms of the number of participants who reported local and systemic reactions up to 6 days after each vaccination per vaccination group.
Time Frame: Up to 6 days after each vaccination.
Population: The analysis was performed on the Safety Set population.
Measure: Number; unit: Participants
Arm/Group | TIV + aH5N1 (18-60 Yrs) | PL+ aTIV (18-60 Yrs)
Number analyzed (Participants) | 2611 | 658
Participants
  Local reactions | 1755 | 502
  Injection site ecchymosis | 237 | 78
  Injection site erythema | 652 | 206
  Injection site induration | 549 | 181
  Injection site swelling | 409 | 162
  Injection site pain | 1537 | 448
  Systemic reactions | 1387 | 386
  Chills | 342 | 118
  Malaise | 347 | 130
  Myalgia | 869 | 277
  Arthralgia | 188 | 79
  Nausea | 193 | 64
  Headache | 668 | 189
  Sweating | 237 | 658
  Fatigue | 638 | 188
  Fever ≥ 38°C | 28 | 12
  Stayed at home | 64 | 22
  Analgesic Antipyretic medi. used | 361 | 114

2. Secondary Outcome: The Number of Subjects With at Least One Reactogenicity Sign After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine as Compared With the Adjuvanted Seasonal Trivalent Influenza Vaccine aTIV.
Description: To evaluate the safety and tolerability profile of two doses of the adjuvanted pandemic H5N1 vaccine (aH5N1) as compared with the MF59-adjuvanted seasonal trivalent influenza vaccine (aTIV), in terms of the number of subjects who reported local and systemic reactions up to 6 days after each vaccination per vaccination group.
Time Frame: Up to 6 days after each vaccination.
Population: The analysis was performed on the Safety set population.
Measure: Number; unit: Subjects
Arm/Group | TIV + aH5N1 (18-60 Yrs) | PL+ aTIV (18-60 Yrs) | TIV + aH5N1 (>60 Yrs) | PL+ aTIV (>60 Yrs)
Number analyzed (Participants) | 2611 | 658 | 214 | 54
Subjects
  Local reactions | 1755 | 502 | 115 | 30
  Injection site ecchymosis (N= 2610,658,214,54): number analyzed (Participants) | 2610 | 658 | 214 | 54
  Injection site ecchymosis (N= 2610,658,214,54) | 237 | 78 | 23 | 7
  Injection site erythema | 652 | 206 | 45 | 14
  Injection site induration (N= 2610,658,214,54): number analyzed (Participants) | 2610 | 658 | 214 | 54
  Injection site induration (N= 2610,658,214,54) | 549 | 181 | 22 | 10
  Injection site swelling | 409 | 162 | 22 | 6
  Injection site pain (N= 2610,658,214,54): number analyzed (Participants) | 2610 | 658 | 214 | 54
  Injection site pain (N= 2610,658,214,54) | 1537 | 448 | 87 | 21
  Systemic reactions | 1387 | 386 | 95 | 26
  Chills | 342 | 118 | 29 | 10
  Malaise (N= 2610,658,214,54): number analyzed (Participants) | 2610 | 658 | 214 | 54
  Malaise (N= 2610,658,214,54) | 347 | 130 | 25 | 6
  Myalgia | 869 | 277 | 59 | 16
  Arthralgia (N= 2610,658,214,54): number analyzed (Participants) | 2610 | 658 | 214 | 54
  Arthralgia (N= 2610,658,214,54) | 188 | 79 | 15 | 5
  Nausea | 193 | 64 | 14 | 3
  Headache (N= 2610,658,214,54): number analyzed (Participants) | 2610 | 658 | 214 | 54
  Headache (N= 2610,658,214,54) | 668 | 189 | 38 | 10
  Sweating | 237 | 63 | 10 | 2
  Fatigue (N= 2610,658,214,54): number analyzed (Participants) | 2610 | 658 | 214 | 54
  Fatigue (N= 2610,658,214,54) | 638 | 188 | 27 | 7
  Fever ≥38°C | 28 | 12 | 1 | 1
  Stayed at home: number analyzed (Participants) | 2591 | 651 | 214 | 54
  Stayed at home | 64 | 22 | 3 | 1
  Analg. Antipyr. Medi. used: number analyzed (Participants) | 2608 | 658 | 214 | 54
  Analg. Antipyr. Medi. used | 361 | 114 | 27 | 6

3. Secondary Outcome: Geometric Mean Titers (GMTs) After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Homologous A/Vietnam/1194/2004 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic H5N1 vaccine (aH5N1), each containing 7.5µg of H5N1 antigen, in terms of GMTs against the homologous A/Vietnam/1194/2004 strain, as determined by Hemagglutination Inhibition (HI) assay and Microneutralization (MN) assay.
Time Frame: Day 22, Day 43, Day 64
Population: The analysis was performed on the Full Analysis Set (FAS) of the Immunogenicity Subset - All subjects in the enrolled population who were in the immunogenicity subset and who actually received at least one dose of AdjPanH5N1 or Adj Seasonal, and provided at leatr one evaluable serum sample both before and after baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- TIV + aH5N1 (18-60 Yrs) HI Assay; TIV + aH5N1 (>60 Yrs) HI Assay; TIV + aH5N1 (18-60 Yrs) MN Assay; TIV + aH5N1 (>60 Yrs) MN Assay: First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1)
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Assay | TIV + aH5N1 (>60 Yrs) HI Assay | TIV + aH5N1 (18-60 Yrs) MN Assay | TIV + aH5N1 (>60 Yrs) MN Assay
Number analyzed (Participants) | 196 | 205 | 197 | 209
Titers
  Day 22 (baseline) | 6.17 [5.58 to 6.83] | 6.98 [6.21 to 7.85] | 11 [10 to 11] | 10 [9.97 to 11]
  Day 43: number analyzed (Participants) | 196 | 201 | 197 | 207
  Day 43 | 14 [11 to 17] | 15 [12 to 18] | 17 [15 to 19] | 17 [15 to 19]
  Day 64: number analyzed (Participants) | 195 | 203 | 197 | 208
  Day 64 | 44 [34 to 56] | 36 [28 to 45] | 65 [56 to 77] | 45 [39 to 53]

4. Secondary Outcome: Geometric Mean Areas (GMAs) After Two Doses of the Adjuvanted Pandemic Vaccine (aH5N1).
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, in terms of GMAs as determined by Single Radial Hemolysis (SRH) assay.
  GMA: For each vaccine group, least squares GMAs (for SRH data), associated 2-sided 95% confidence interval and median, minimal, and maximal titer values were determined for study Day 22, Day 43 and Day 64.
Time Frame: Day 22, Day 43, Day 64
Population: The analysis was performed on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: Areas (mm^2)
Groups:
- TIV + aH5N1 (>60 Yrs): First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) | TIV + aH5N1 (>60 Yrs)
Number analyzed (Participants) | 197 | 210
Areas (mm^2)
  Day 22 (baseline) | 11 [9.45 to 12] | 13 [11 to 14]
  Day 43: number analyzed (Participants) | 197 | 208
  Day 43 | 21 [18 to 24] | 20 [18 to 23]
  Day 64: number analyzed (Participants) | 197 | 209
  Day 64 | 43 [39 to 47] | 37 [33 to 41]

5. Secondary Outcome: Geometric Mean Ratios (GMRs) After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Homologous A/Vietnam/1194/2004 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine (aH5N1), each containing 7.5µg of H5N1 antigen,in terms of GMRs against the homologous A/Vietnam/1194/2004 strain, as determined by HI, MN and SRH assays.
Time Frame: Day 43/Day 22, Day 64/Day 22
Population: The analysis was performed on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Groups:
- TIV + aH5N1 (18-60 Yrs) HI Assay; TIV + aH5N1 (>60 Yrs) HI Assay; TIV + aH5N1 (18-60 Yrs) MN Assay; TIV + aH5N1 (>60 Yrs) MN Assay: First dose of the non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of the adjuvanted pandemic H5N1 vaccine (aH5N1).
- TIV + aH5N1 (18-60 Yrs) SRH Assay; TIV + aH5N1 (>60 Yrs) SRH Assay: First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Assay | TIV + aH5N1 (>60 Yrs) HI Assay | TIV + aH5N1 (18-60 Yrs) MN Assay | TIV + aH5N1 (>60 Yrs) MN Assay | TIV + aH5N1 (18-60 Yrs) SRH Assay | TIV + aH5N1 (>60 Yrs) SRH Assay
Number analyzed (Participants) | 196 | 203 | 197 | 208 | 197 | 209
Ratios
  Day 43 to Day 22 (N= 196,201,197,207,197,208): number analyzed (Participants) | 196 | 201 | 197 | 207 | 197 | 208
  Day 43 to Day 22 (N= 196,201,197,207,197,208) | 2.25 [1.86 to 2.72] | 2.14 [1.8 to 2.54] | 1.58 [1.39 to 1.79] | 1.63 [1.43 to 1.84] | 1.95 [1.72 to 2.2] | 1.57 [1.41 to 1.75]
  Day 64 to Day 22: number analyzed (Participants) | 195 | 203 | 197 | 208 | 197 | 209
  Day 64 to Day 22 | 7.1 [5.52 to 9.14] | 5.15 [4.15 to 6.4] | 6.21 [5.29 to 7.29] | 4.42 [3.79 to 5.15] | 4.03 [3.54 to 4.59] | 2.9 [2.53 to 3.31]

6. Secondary Outcome: Percentages of Subjects With HI Titers ≥ 40 and GMAs ≥ 25mm^2, After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Homologous A/Vietnam/1194/2004 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, each containing 7.5µg of H5N1 antigen, against the homologous A/Vietnam/1194/2004 strain, in terms of percentages of subjects achieving HI titers ≥ 40 and GMAs ≥ 25mm^2, as determined by HI and SRH assays.
  GMA: For each vaccine group, least squares GMAs (for SRH data), associated 2-sided 95% confidence interval and median, minimal, and maximal titer values were determined for study Day 22, Day 43 and Day 64.
Time Frame: Day 22, Day 43 and Day 64
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- TIV + aH5N1 (18-60 Yrs) HI Titers ≥ 40; TIV + aH5N1 (>60 Yrs) HI Titers ≥ 40; TIV + aH5N1 (>60 Yrs) SRH Areas ≥ 25mm^2: First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
- TIV + H5N1 (18-60 Yrs) SRH Areas ≥ 25mm^2: First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Titers ≥ 40 | TIV + aH5N1 (>60 Yrs) HI Titers ≥ 40 | TIV + H5N1 (18-60 Yrs) SRH Areas ≥ 25mm^2 | TIV + aH5N1 (>60 Yrs) SRH Areas ≥ 25mm^2
Number analyzed (Participants) | 196 | 205 | 197 | 210
Percentages of subjects
  Day 22 (baseline) | 6 [3 to 10] | 8 [5 to 12] | 19 [14 to 26] | 25 [20 to 32]
  Day 43: number analyzed (Participants) | 196 | 201 | 197 | 208
  Day 43 | 30 [23 to 37] | 31 [25 to 38] | 48 [41 to 55] | 46 [39 to 53]
  Day 64: number analyzed (Participants) | 195 | 203 | 197 | 209
  Day 64 | 61 [53 to 67] | 57 [50 to 64] | 91 [87 to 95] | 82 [76 to 87]

7. Secondary Outcome: Percentages of Subjects Achieving Seroconversion or Significant Increase in Antibody Titer After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Homologous A/Vietnam/1194/2004 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, each containing 7.5µg of H5N1 antigen, against the homologous A/Vietnam/1194/2004 strain, in terms of percentages of subjects achieving seroconversion or significant increase in antibody titer as measured by HI and SRH assays.
Time Frame: Day 43/Day 22 and Day 64/Day 22
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- TIV + aH5N1 (18-60 Yrs) HI Titers; TIV + aH5N1 (18-60 Yrs) SRH Areas; TIV + aH5N1 (>60 Yrs) SRH Areas: First dose of the non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of the adjuvanted pandemic H5N1 vaccine (aH5N1).
- TIV + aH5N1 (>60 Yrs) HI Titers: First dose of the non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of the adjuvanted pandemic H5N1 vaccine (H5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Titers | TIV + aH5N1 (>60 Yrs) HI Titers | TIV + aH5N1 (18-60 Yrs) SRH Areas | TIV + aH5N1 (>60 Yrs) SRH Areas
Number analyzed (Participants) | 196 | 203 | 197 | 209
Percentages of subjects
  Day 43/Day 22: number analyzed (Participants) | 196 | 201 | 197 | 208
  Day 43/Day 22 | 23 [18 to 30] | 22 [16 to 28] | 37 [30 to 44] | 23 [17 to 29]
  Day 64/Day 22: number analyzed (Participants) | 195 | 203 | 197 | 208
  Day 64/Day 22 | 56 [49 to 63] | 50 [43 to 57] | 78 [72 to 84] | 63 [56 to 69]

8. Secondary Outcome: GMTs After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Heterologous A/Turkey/Turkey/1/2005 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine (aH5N1), each containing 7.5µg of H5N1 antigen, in terms of GMTs against the heterologous A/turkey/Turkey/1/2005 strain, as determined by HI and MN assays.
Time Frame: Day 22, Day 43 and Day 64
Population: The analysis was performed on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- TIV + aH5N1 (>60 Yrs) HI Assay: First dose of non-adjuvanted seasonal trivalent influenza vaccine (eTIV_a) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Assay | TIV + aH5N1 (>60 Yrs) HI Assay | TIV + aH5N1 (18-60 Yrs) MN Assay | TIV + aH5N1 (>60 Yrs) MN Assay
Number analyzed (Participants) | 197 | 208 | 197 | 210
Titers
  Day 22 (baseline) | 6.03 [5.55 to 6.55] | 6.85 [6.21 to 7.55] | 11 [10 to 11] | 11 [11 to 12]
  Day 43: number analyzed (Participants) | 197 | 206 | 196 | 207
  Day 43 | 8.03 [7.07 to 9.12] | 8.87 [7.69 to 10] | 15 [13 to 17] | 15 [13 to 16]
  Day 64: number analyzed (Participants) | 197 | 207 | 197 | 208
  Day 64 | 12 [9.77 to 14] | 12 [10 to 14] | 30 [26 to 35] | 23 [20 to 26]

9. Secondary Outcome: GMAs After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Heterologous A/Turkey/Turkey/1/2005 Strain.
Description: To evaluate the immunogenicity of two doses of adjuvanted pandemic vaccine aH5N1, each containing 7.5µg of H5N1 antigen, in terms of GMAs against the heterologous A/turkey/Turkey/1/2005 strain, as determined by SRH assay.
  GMA: For each vaccine group, least squares GMAs (for SRH data), associated 2-sided 95% confidence interval and median, minimal, and maximal titer values were determined for study Day 22, Day 43 and Day 64.
Time Frame: Day 22, Day 43 and Day 64
Population: The analysis was performed on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: Areas (mm^2)
Groups:
- TIV + aH5N1 (18-60 Yrs); TIV + aH5N1 (>60 Yrs): First dose of the non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of the adjuvanted pandemic H5N1 vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) | TIV + aH5N1 (>60 Yrs)
Number analyzed (Participants) | 197 | 210
Areas (mm^2)
  Day 22 (baseline) | 9.89 [8.82 to 11] | 12 [10 to 13]
  Day 43: number analyzed (Participants) | 196 | 208
  Day 43 | 14 [13 to 16] | 14 [13 to 16]
  Day 64: number analyzed (Participants) | 197 | 209
  Day 64 | 23 [21 to 26] | 20 [18 to 23]

10. Secondary Outcome: GMRs After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Heterologous A/Turkey/Turkey/1/2005 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, each containing 7.5µg of H5N1 antigen, in terms of GMRs against the heterologous A/turkey/Turkey/1/2005 strain, as determined by HI, MN and SRH assays.
Time Frame: Day 43/Day 22 and Day 64/Day 22
Population: The analysis was performed on FAS population.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Groups:
- TIV + aH5N1 (18-60 Yrs) SRH Assay; TIV + aH5N1 (>60 Yrs) SRH Assay: First dose of the non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of the adjuvanted pandemic H5N1 vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Assay | TIV + aH5N1 (>60 Yrs) HI Assay | TIV + aH5N1 (18-60 Yrs) MN Assay | TIV + aH5N1 (>60 Yrs) MN Assay | TIV + aH5N1 (18-60 Yrs) SRH Assay | TIV + aH5N1 (>60 Yrs) SRH Assay
Number analyzed (Participants) | 197 | 207 | 197 | 208 | 197 | 209
Ratios
  Day 43/Day 22 | 1.33 [1.19 to 1.49] | 1.29 [1.16 to 1.45] | 1.39 [1.25 to 1.54] | 1.29 [1.17 to 1.42] | 1.44 [1.31 to 1.59] | 1.25 [1.15 to 1.36]
  Day 64/Day 22 | 1.92 [1.64 to 2.25] | 1.79 [1.56 to 2.06] | 2.77 [2.4 to 3.2] | 2.01 [1.78 to 2.26] | 2.37 [2.1 to 2.67] | 1.74 [1.57 to 1.94]

11. Secondary Outcome: Percentages of Subjects With HI ≥ 40 and GMAs ≥ 25mm^2, After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Heterologous A/Turkey/Turkey/1/2005 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, each containing 7.5µg of H5N1 antigen, against the heterologous A/turkey/Turkey/1/2005 strain, in terms of percentages of subjects achieving HI titers ≥ 40 and GMAs ≥ 25mm^2 as determined by HI and SRH assays.
  GMA: For each vaccine group, least squares GMAs (for SRH data), associated 2-sided 95% confidence interval and median, minimal, and maximal titer values were determined for study Vaccine on Day 22, Day 43, Day 64.
Time Frame: Day 22, Day 43 and Day 64
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- TIV + aH5N1 (18-60 Yrs) SRH Areas ≥ 25mm^2; TIV + aH5N1 (>60 Yrs) SRH Areas≥ 25mm^2: First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Titers ≥ 40 | TIV + aH5N1 (>60 Yrs) HI Titers ≥ 40 | TIV + aH5N1 (18-60 Yrs) SRH Areas ≥ 25mm^2 | TIV + aH5N1 (>60 Yrs) SRH Areas≥ 25mm^2
Number analyzed (Participants) | 197 | 208 | 197 | 210
Percentages of subjects
  Day 22 (baseline) | 3 [1 to 7] | 5 [2 to 9] | 16 [11 to 22] | 23 [18 to 30]
  Day 43: number analyzed (Participants) | 197 | 206 | 196 | 208
  Day 43 | 11 [7 to 16] | 15 [10 to 20] | 30 [24 to 37] | 32 [26 to 39]
  Day 64: number analyzed (Participants) | 197 | 207 | 197 | 209
  Day 64 | 23 [18 to 30] | 25 [19 to 32] | 59 [52 to 66] | 48 [41 to 55]

12. Secondary Outcome: Percentages of Subjects Achieving Seroconversion or Significant Increase in Antibody Titers, After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Heterologous A/Turkey/Turkey/1/2005 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, each containing 7.5µg of H5N1 antigen, against the heterologous A/turkey/Turkey/1/2005 strain, in terms of percentages of subjects achieving seroconversion or significant increase in antibody titer as measured by HI and SRH assays.
Time Frame: Day 43/Day 22 and Day 64/Day 22)
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- TIV + aH5N1 (18-60 Yrs) HI Titers; TIV + aH5N1 (>60 Yrs) HI Titers; TIV + aH5N1 (18-60 Yrs) SRH Areas; TIV + aH5N1 (>60 Yrs) SRH Areas: First dose of non-adjuvanted seasonal trivalent influenza vaccine (TIV) followed by two doses of adjuvanted pandemic H5N1 vaccine (aH5N1).
Arm/Group | TIV + aH5N1 (18-60 Yrs) HI Titers | TIV + aH5N1 (>60 Yrs) HI Titers | TIV + aH5N1 (18-60 Yrs) SRH Areas | TIV + aH5N1 (>60 Yrs) SRH Areas
Number analyzed (Participants) | 197 | 207 | 197 | 209
Percentages of subjects
  Day 43/Day 22 | 9 [5 to 13] | 8 [5 to 12] | 18 [13 to 24] | 10 [6 to 14]
  Day 64/Day 22 | 19 [14 to 25] | 19 [14 to 25] | 49 [42 to 56] | 32 [26 to 39]

13. Primary Outcome: Number of Subjects Exposed to Adjuvanted Pandemic Influenza Vaccine.
Description: To report safety data from a large enough number of subjects exposed to adjuvanted pandemic influenza vaccine aH5N1 capable of detecting rare adverse events (AEs), i.e. events occurring at a frequency of <=0.1%, & uncommon AEs in elderly, i.e. occurring at a frequency of <=1% of subjects.
Time Frame: Upto Day 224 post vaccination
Population: The analysis was performed on the Safety set population.
Measure: Number; unit: Participants
Arm/Group | TIV + aH5N1 (18-60 Yrs) | PL+ aTIV (18-60 Yrs) | TIV + aH5N1 (>60 Yrs) | PL+ aTIV (>60 Yrs)
Number analyzed (Participants) | 2693 | 679 | 219 | 56
Participants | 2692 | 679 | 219 | 56

14. Secondary Outcome: Percentages of Subjects With MN Titers ≥20, ≥40, ≥80, After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Homologous A/Vietnam/1194/2004 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine (aH5N1), each containing 7.5μg of H5N1 antigen, against the homologous A/Vietnam/1194/2004 strain, in terms of percentages of subjects achieving MN Titers ≥20, ≥ 40, ≥80 on Days 22, Day 43 and Day 64.
Time Frame: Day 22, Day 43 and Day 64
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV + aH5N1 (18-60 Yrs) | TIV + aH5N1 (>60 Yrs)
Number analyzed (Participants) | 197 | 209
Percentages of subjects
  Day 22 (MN titer ≥ 20) | 3 [1 to 6] | 2 [1 to 5]
  Day 43 (MN titer ≥ 20): number analyzed (Participants) | 197 | 207
  Day 43 (MN titer ≥ 20) | 27 [21 to 34] | 25 [19 to 31]
  Day 64 (MN titer ≥ 20): number analyzed (Participants) | 197 | 208
  Day 64 (MN titer ≥ 20) | 79 [73 to 85] | 72 [65 to 78]
  Day 22 (MN titer ≥ 40) | 2 [0 to 4] | 1 [0 to 3]
  Day 43 (MN titer ≥ 40): number analyzed (Participants) | 197 | 207
  Day 43 (MN titer ≥ 40) | 16 [11 to 22] | 19 [14 to 25]
  Day 64 (MN titer ≥ 40): number analyzed (Participants) | 197 | 208
  Day 64 (MN titer ≥ 40) | 67 [60 to 74] | 57 [50 to 64]
  Day 22 (MN titer ≥ 80) | 1 [0 to 4] | 0 [0 to 2]
  Day 43 (MN titer ≥ 80): number analyzed (Participants) | 197 | 207
  Day 43 (MN titer ≥ 80) | 9 [6 to 14] | 13 [8 to 18]
  Day 64 (MN titer ≥ 80): number analyzed (Participants) | 197 | 208
  Day 64 (MN titer ≥ 80) | 50 [43 to 57] | 33 [26 to 40]

15. Secondary Outcome: Percentages of Subjects With MN Titers ≥20, ≥40, ≥80, After Two Doses of the Adjuvanted Pandemic aH5N1 Vaccine Against the Heterologous A/Turkey/Turkey/1/2005 Strain.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, each containing 7.5μg of H5N1 antigen, against the heterologous A/turkey/Turkey/1/2005 Strain, in terms of percentages of subjects achieving MN Titers ≥20, ≥ 40, ≥80 on Day 22, Day 43 and Day 64.
Time Frame: Day 22, Day 43 and Day 64
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV + aH5N1 (18-60 Yrs) | TIV + aH5N1 (>60 Yrs)
Number analyzed (Participants) | 197 | 210
Percentages of subjects
  Day 22 (MN titer≥20) | 5 [2 to 8] | 9 [6 to 14]
  Day 43 (MN titer ≥ 20): number analyzed (Participants) | 196 | 207
  Day 43 (MN titer ≥ 20) | 23 [17 to 29] | 21 [15 to 27]
  Day 64 (MN titer ≥ 20; N= 197, 208): number analyzed (Participants) | 197 | 208
  Day 64 (MN titer ≥ 20; N= 197, 208) | 59 [52 to 66] | 47 [40 to 54]
  Day 22 (MN titer ≥ 40) | 3 [1 to 7] | 3 [1 to 7]
  Day 43 (MN titer ≥ 40): number analyzed (Participants) | 196 | 208
  Day 43 (MN titer ≥ 40) | 13 [8 to 18] | 14 [9 to 19]
  Day 64 (MN titer ≥ 40): number analyzed (Participants) | 197 | 208
  Day 64 (MN titer ≥ 40) | 39 [32 to 46] | 30 [24 to 37]
  Day 22 (MN titer ≥ 80) | 2 [1 to 5] | 0.012 [0.012 to 3]
  Day 43 (MN titer ≥ 80): number analyzed (Participants) | 196 | 207
  Day 43 (MN titer ≥ 80) | 8 [4 to 12] | 6 [3 to 10]
  Day 64 (MN titer ≥ 80): number analyzed (Participants) | 197 | 208
  Day 64 (MN titer ≥ 80) | 19 [14 to 26] | 12 [8 to 17]

16. Secondary Outcome: Percentages of Subjects Achieving at Least a Four-fold Rise in MN Antibody Titer on Day 43 and Day 64, Compared to Day 22 Against Homologous Strains.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine aH5N1, each containing 7.5μg of H5N1 antigen, against the homologous A/Vietnam/1194/2004 strain, in terms of percentages of subjects achieving at least a four-fold rise in MN antibody titer on Day 43 and Day 64, compared to Day 22.
Time Frame: Day 43/Day 22 and Day 64/Day 22
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV + aH5N1 (18-60 Yrs) | TIV + aH5N1 (>60 Yrs)
Number analyzed (Participants) | 197 | 208
Percentages of subjects
  Day 43/Day 22: number analyzed (Participants) | 197 | 207
  Day 43/Day 22 | 14 [10 to 20] | 18 [13 to 24]
  Day 64/Day 22 | 65 [58 to 72] | 55 [48 to 62]

17. Secondary Outcome: Percentages of Subjects Achieving at Least a Four-fold Rise in MN Antibody Titer on Day 43 and Day 64, Compared to Day 22 Against Heterologous Strains.
Description: To evaluate the immunogenicity of two doses of the adjuvanted pandemic vaccine (aH5N1), each containing 7.5μg of H5N1 antigen, against Heterologous A/turkey/Turkey/1/2005 Strain, in terms of percentages of subjects achieving at least a four-fold rise in MN antibody titer on Day 43 and Day 64, compared to Day 22.
Time Frame: Day 43/Day 22 and Day 64/Day 22
Population: The analysis was performed on FAS population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | TIV + aH5N1 (18-60 Yrs) | TIV + aH5N1 (>60 Yrs)
Number analyzed (Participants) | 197 | 208
Percentages of subjects
  Day 43/Day 22: number analyzed (Participants) | 196 | 207
  Day 43/Day 22 | 9 [5 to 14] | 9 [6 to 14]
  Day 64/Day 22 | 36 [29 to 43] | 25 [19 to 31]

18. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs After Vaccination.
Description: The number of subjects reporting any unsolicited AEs any, Possibly/probably related AEs, serious adverse events (SAEs), AEs leading to withdrawal (WD), AEs leading to death from Day 1 through Day 224 post vaccination.
Time Frame: Day 1 through Day 224 post vaccination
Population: Analysis was done on safety population.
Measure: Number; unit: Subjects
Groups:
- PL + aTIV (18-60 Yrs); PL + aTIV (>60 Yrs): First dose of placebo (PL) followed by two doses of adjuvanted seasonal trivalent influenza vaccine (aTIV).
Arm/Group | TIV + aH5N1 (18-60 Yrs) | PL + aTIV (18-60 Yrs) | TIV + aH5N1 (>60 Yrs) | PL + aTIV (>60 Yrs)
Number analyzed (Participants) | 2611 | 658 | 214 | 54
Subjects
  Any AEs | 1329 | 335 | 103 | 29
  SAEs | 45 | 10 | 4 | 3
  At least possibly related AEs | 357 | 103 | 25 | 13
  AEs Leading to Premature Withdrawal | 4 | 4 | 2 | 1
  Deaths | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study ie. Day 1 to Day 224
Description: The number of subjects in the module for Adverse Events (AEs) differs from the number of subjects in the Participant Flow module. This is because the analysis for the AEs module is based on the safety population whereas the Participant Flow module refers to the enrolled population.
Arm/Group | TIV + aH5N1 (18-60 Yrs) | PL + aTIV (18-60 Yrs) | TIV + aH5N1 (>60 Yrs) | PL + aTIV (>60 Yrs)
Serious Adverse Events (participants affected / at risk) | 40/2680 | 9/676 | 1/222 | 2/56
Other Adverse Events (participants affected / at risk) | 2301/2680 | 590/676 | 176/222 | 45/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIV + aH5N1 (18-60 Yrs) (N=2680) | PL + aTIV (18-60 Yrs) (N=676) | TIV + aH5N1 (>60 Yrs) (N=222) | PL + aTIV (>60 Yrs) (N=56)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster opthalmic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gas poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebellar haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infraction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia,paranoid type (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral caruncle (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial hyperactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIV + aH5N1 (18-60 Yrs) (N=2680) | PL + aTIV (18-60 Yrs) (N=676) | TIV + aH5N1 (>60 Yrs) (N=222) | PL + aTIV (>60 Yrs) (N=56)
Nausea (Gastrointestinal disorders) | 334 (334) | 88 (88) | 19 (19) | 4 (4)
Chills (General disorders) | 532 (532) | 152 (152) | 40 (40) | 13 (13)
Fatigue (General disorders) | 927 (927) | 247 (247) | 38 (38) | 9 (9)
Injection site erythema (General disorders) | 1041 (1041) | 248 (248) | 87 (87) | 18 (18)
Injection site haemorrahage (General disorders) | 367 (367) | 111 (111) | 33 (33) | 13 (13)
Injection site induration (General disorders) | 830 (830) | 195 (195) | 42 (42) | 13 (13)
Injection site pain (General disorders) | 1738 (1738) | 459 (459) | 96 (96) | 21 (21)
Injection site swelling (General disorders) | 632 (632) | 177 (177) | 28 (28) | 6 (6)
Malaise (General disorders) | 542 (542) | 161 (161) | 33 (33) | 7 (7)
Nasopharyngitis (Infections and infestations) | 216 (216) | 59 (59) | 7 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 176 (176) | 44 (44) | 8 (8) | 5 (5)
Rhinitis (Infections and infestations) | 83 (83) | 27 (27) | 4 (4) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 306 (306) | 97 (97) | 19 (19) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1088 (1088) | 296 (296) | 69 (69) | 17 (17)
Headache (Nervous system disorders) | 1031 (1031) | 253 (253) | 54 (54) | 18 (18)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 356 (356) | 84 (84) | 14 (14) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less